CLINICAL TRIAL: NCT03471442
Title: Erector Spinae Plane Block Versus Paravertebral Block in Patients Undergoing Elective Breast Surgery. A Randomized Controlled Trial Comparing Dermatomal Spread.
Brief Title: Erector Spinae Plane Block Versus Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00078230
Record Dates: First submitted 2018-03-01; First posted 2018-03-20 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Pain, Postoperative; Anesthesia, Local
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Anesthetics, General; Analgesics, Opioid; Anesthetics, Local; Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral (Active Comparator): Ultrasound-guided paravertebral block performed pre-operatively with 20ml of a ropivacaine / bupivacaine mixture.
  Interventions: Procedure: Paravertebral block; Drug: General anesthetic; Drug: Opioids; Drug: Anesthetics, Local
- Erector spinae plane (Experimental): Ultrasound-guided erector spinae plane block performed pre-operatively with 20ml of a ropivacaine / bupivacaine mixture.
  Interventions: Procedure: Erector spinae plane block; Drug: General anesthetic; Drug: Opioids; Drug: Anesthetics, Local

INTERVENTIONS:
Procedure: Paravertebral block — Ultrasound-guided paravertebral block performed pre-operatively in the anesthesia block room with 20ml of a ropivacaine / bupivacaine mixture.
  Arms: Paravertebral
Procedure: Erector spinae plane block — Ultrasound-guided erector spinae plane block performed pre-operatively in the anesthesia block room with 20ml of a ropivacaine / bupivacaine mixture.
  Arms: Erector spinae plane
Drug: General anesthetic — General anesthesia administered as per preference of intra-operative attending anesthesiologist
Drug: Opioids — Intra-operatively, opioids will be titrated to heart rate and spontaneous respiration rate e.g. fentanyl, morphine, hydromorphone. Post-operatively in post anesthesia care unit, morphine and hydromorphone will be titrated to effect as necessary. After discharge from post anesthesia care unit, oral analgesia will be administered on an as required basis e.g. acetaminophen, non-steroid anti-inflammatory medications, acetaminophen / codeine and acetaminophen / oxycodone.
Drug: Anesthetics, Local — Weight-based dosing of this local anesthetic mixture.
  Other Names: Ropivacaine / bupivacaine mixture to a final concentration of 0.125% bupivacaine and 0.5% ropivacaine

SUMMARY:
This study aims to compare the effectiveness of paravertebral block and erector spinae plane block after mastectomy.

The primary objective of this randomized controlled trial is to demonstrate equivalent dermatomal spread for ultrasound-guided single-injection Erector Spinae Plane (ESP) block performed at T4-T5 level and ultrasound-guided single-injection (paravertebral) PVB block at the same level.

Secondary objectives are Numerical Rating Scale (NRS) pain scores in the first 24 post-operative hours, opioid analgesia use intra-operatively and in the first 24 post-operative hours, block procedural time and patient discomfort during block insertion.

The investigators hypothesize that ESP block efficacy is not inferior to PVB with reference to dermatomal sensory spread and analgesic efficacy, while being easier to perform with less associated discomfort during block insertion.

DETAILED DESCRIPTION:
Paravertebral block (PVB) has been shown to provide excellent analgesia for major breast surgery. Advantages of a PVB technique include reduced postoperative pain, analgesic consumption, opioid-related side effects, and shorter post anesthesia care unit (PACU) stay. There is also evidence to suggest that PVB may have a favorable impact on cancer recurrence after mastectomy. Paravertebral blockade results in somatosensory and sympathetic blockade after injection of local anesthetic solution to the paravertebral space posterior to the pleura. Erector spinae plane (ESP) block is a recently described technique which may be an alternative to PVB for providing thoracic analgesia. Numerous case reports and case series describe ESP block for the management of acute and chronic thoracic pain. It involves injection of local anesthetic into the fascial plane deep to erector spinae muscle. Radiological imaging in a cadaver model has demonstrated that a single injection at the level of the T5 transverse process produced cranio-caudal spread between C7 and T8. This accounts for the extensive sensory block that has been observed in case reports and is at least as extensive as the spread seen with PVB.

ESP is a more superficial block with a better defined end-point - injection between the bony transverse process and erector spinae muscle. A more superficial ultrasound-guided block will be faster to perform and less painful for the patient. Furthermore, ESP does not have the same risk of pneumothorax as PVB.There have been no randomized controlled trials involving ESP to date. All descriptions of the technique have been in case report / series format.

The investigators hypothesize that ESP block efficacy is not inferior to PVB with reference to dermatomal sensory spread and analgesic efficacy, while being easier to perform, has less associated discomfort and fewer complication risks.

All eligible participants will be randomized to the PVB arm or the ESP arm after fully informed consent has been obtained. Subjects randomized to the PVB arm will have an ultrasound-guided paravertebral block performed pre-operatively in the anesthesia block room with 20ml of a ropivacaine / bupivacaine mixture. Subjects randomized to the ESP arm will have an ultrasound-guided erector spinae plane block performed pre-operatively in the anesthesia block room with 20ml of a ropivacaine / bupivacaine mixture. Conduct of intra-operative anesthesia will be at the discretion of the attending anesthesiologist.

The primary outcome is equivalent dermatomal spread for ultrasound-guided single-injection ESP block performed at T4-T5 level and ultrasound-guided single-injection PVB block at the same level.

Secondary outcomes are NRS pain scores in the first 24 post-operative hours, opioid analgesia use intra-operatively and in the first 24 post-operative hours, block procedural time and patient discomfort during block insertion.

The primary outcome will be collected by a research associate who is blinded to the study group allocation. The secondary outcomes will be collected by the study team from the patient chart and through patient interview. Continuous variables will be analyzed using t-tests and categorical variables will be analyzed using chi-squared test. Markers of intervention safety will be monitored included local anesthetic toxicity, nerve injury, infection and pneumothorax.

A test of equivalence will be performed for the primary outcome of dermatomal spread between the 2 groups. If the equivalence is not established for the block extent, a 2-way superiority will be conducted. Secondary outcomes will be analyzed using Mann-Whitney U test and the Hodges-Lehmann method for calculating 95% confidence intervals (CIs) around the median difference. Assuming a median difference of 1.5 dermatomal segments, and a pooled standard deviation (SD) of 1.65 segments, α of 0.05, and 90% power, a total sample size of 42 patients is estimated (21 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years
* Consented to a regional anesthesia technique for post-operative analgesia
* Partial or complete mastectomy

Exclusion Criteria:

* Subjects <18 years
* those who refuse consent for PVB or ESP blockade,
* opioid tolerant patients
* psychiatric illness
* allergy to local anesthetic
* Local or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Dermatomal spread of sensory blockade | 30 minutes
  Assessment of extent of sensory block by pinprick

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for pain | Up to 24 hours
  Subjective pain score between 0 (no pain) and 10 (worst possible pain) immediately post-operatively at 6, 12 and 24 hours
Opioid analgesia use intra-operatively | 1 to 3 hours
  Amount of opioid administered by the intra-operative anesthesiologist
Total opioid use in the first 24 hours | Up to 24 hours
  Amount of opioid used by patient in the first 24 hours after surgery
Block procedural time | Up to 30 Minutes
  Amount of time it takes to perform the block procedure starting with when the ultrasound image is acquired and finishing when all of the local anesthetic has been injected

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boughey JC, Goravanchi F, Parris RN, Kee SS, Frenzel JC, Hunt KK, Ames FC, Kuerer HM, Lucci A. Improved postoperative pain control using thoracic paravertebral block for breast operations. Breast J. 2009 Sep-Oct;15(5):483-8. doi: 10.1111/j.1524-4741.2009.00763.x. Epub 2009 Jul 13. PMID 19624418
- [Background] Abdallah FW, Morgan PJ, Cil T, McNaught A, Escallon JM, Semple JL, Wu W, Chan VW. Ultrasound-guided multilevel paravertebral blocks and total intravenous anesthesia improve the quality of recovery after ambulatory breast tumor resection. Anesthesiology. 2014 Mar;120(3):703-13. doi: 10.1097/ALN.0000436117.52143.bc. PMID 24071616
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016